CLINICAL TRIAL: NCT03504384
Title: Cross Cultural Adaptation and Validation of The Arabic Version Of EuroQol 5D-5L
Brief Title: Adaptation and Validation of the Arabic Version of EuroQol 5D-5L
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ahmed Sarhan, dr, Assiut University
Other Study IDs: validation of EuroQol 5D-5L
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Validation Study
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — All patients will be interviewed using a semi-structured questionnaire detailing patients' demographic characteristics (age, sex, education, occupation, residence), and the factors that could affect their quality of life such as pain and neurological symptoms, orthopedic disorder in another part of the body and history of spinal surgery.

SUMMARY:
The aim of the work is to provide a validated Arabic version of EuroQol 5D-5L ,so that it would be used as a quality of life assessment tool for Egyptian patients

Specific objectives:

1. Cross cultural adaptation of the translated Arabic version of EuroQol 5D-5L.
2. Assessment of the reliability of the translated Arabic version of EuroQol 5D-5L.
3. Testing the validity of the translated version of EuroQol 5D-5L.

DETAILED DESCRIPTION:
Chronic back pain is one of the most important disabling illnesses. It has a high incidence, high prevalence and high cost to society. One of the most common causes of back pain are degenerative spine diseases which aﬀect all aspects of quality of life (QoL) of the patients. They could aﬀect job opportunities, social activities and hinder the patients from performing common daily activities.It was found that many factors could affect quality of life of spine degenerative diseases patients such as sex, age, body mass index (BMI), employment status , living with other family members, smoking, orthopedic disorder in another part of the body (other than spinal disease), history of spinal surgery, and bladder function. Comprehensive assessment of these patients should include health related quality of life (HRQoL) measures in addition to the objective clinical measures of the diseases. Europeans Quality of life questionnaire 5 dimensions ,5 levels (EQ-5D-5L) is a standardized measure of health status developed by the EuroQol Group which provides a simple, generic measure of health for clinical and economic appraisal (2).Despite being translated and validated in many languages, there is no validated Arabic version of EQ-5D-5L to measure the quality of life. The objective of this study is to evaluate the reliability and validity of the Arabic version of the questionnaire for Egyptian patients diagnosed to have Spine degenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients operated upon for spine degenerative disease coming for follow up in the outpatient clinics.

Exclusion Criteria:

* preoperative patients and immediate postoperative patients.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: between 18 and 70 years old. patients operated upon for spine degenerative disease coming for follow up in the outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
A reliable and validated Arabic version of the EQ-5D-5L instrument | basline
  Cross cultural adaptation and validation of the Arabic version of the EQ-5D-5L.

SECONDARY OUTCOMES:
factors affecting quality of life of spine disease patients. | baseline
  to study factors affecting quality of life of spine disease patients.

REFERENCES:
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569